CLINICAL TRIAL: NCT03432026
Title: Chronic Obstructive Pulmonary Disease Phenotypes in Non-Smokers
Brief Title: Phenotypes of COPD
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, C F Shamshon, Principal investigator, Assiut University
Other Study IDs: COPD
Record Dates: First submitted 2018-01-22; First posted 2018-02-13 (Actual); Last update posted 2018-06-27 (Actual); Status verified 2018-06

CONDITIONS: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Non-smoker COPD patients: stable non-smoker COPD patients diagnosed by a previous spiromtery to have FEV1/FVC less than 70
  Interventions: Device: High resolution computed tomography scan of the chest.

INTERVENTIONS:
Device: High resolution computed tomography scan of the chest. — High resolution computed tomography scan of the chest & pulmonary function tests will be done for every patient to classify them.

SUMMARY:
Chronic Obstructive Pulmonary Disease (COPD) has been defined by international guidelines as a common preventable and treatable disease characterized by persistent air flow limitation and respiratory symptoms caused by exposure to gases or noxious particles.

COPD is a major cause of morbidity and mortality worldwide. It is predicted to become the third leading cause of death and the fifth leading cause of disability by the year 2020.

DETAILED DESCRIPTION:
Although the disease has been greatly associated with tobacco smoking, non- smokers can also have COPD, and the burden of COPD in non-smokers is also higher than previously believed especially in developing countries. Exposure to gases, environmental pollution, respiratory infection, noxious particles, passive smoking, and indoor air pollution is the main cause of COPD in non smokers.

COPD over the years has been classified into two phenotypes; chronic bronchitis or classic emphysema.However, The Global Initiative for Chronic Obstructive Lung Disease (GOLD) guidelines over the last few years have stopped emphasizing the categorization of chronic obstructive pulmonary disease (COPD) into only emphysema or chronic bronchitis

Clear examples of COPD phenotypes in smokers have been described in different Researches,such as emphysema, chronic bronchitis, frequent exacerbators and the asthma_copd overlap.,but there is alack of information about COPD phenotypes in non-smokers, So, there is a continuous need for research into groups of non smoking patients.

Therefore, the aim of this study is to describe the phenotypes of COPD, their risk factors, Clinical and functional assessment and the prognosis of each COPD phenotype in non-smoking patients.

ELIGIBILITY:
Inclusion Criteria:

1. Non-smoker COPD patients.
2. Stable COPD patients (≥4 weeks without exacerbation or worsening of any relevant comorbidity).

Exclusion Criteria:

1. Patients with COPD exacerbation.
2. Patients with associated obstructive sleep apnea.
3. Patients with associated interstitial lung disease.
4. patients with associated cardiac problems.
5. Patients with associated bronchiaectasis.

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Non smoker COPD stable patients
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2019-04-01 (Estimated); Primary Completion 2020-04-01 (Estimated); Study Completion 2021-04-01 (Estimated)

PRIMARY OUTCOMES:
Rate of risk factors of COPD in non smokers. | 48 hour
  Complete medical history will be taken for each patient to detect risk factors of COPD.

REFERENCES:
- [Background] Sharma BB, Singh V. Nonsmoker COPD: Is it a reality? Lung India. 2017 Mar-Apr;34(2):117-119. doi: 10.4103/lungindia.lungindia_56_17. No abstract available. PMID 28360456
- [Background] Mohan A, Sharma M, Uniyal A, Borah R, Luthra K, Pandey RM, Madan K, Hadda V, Guleria R. Variability in proteinase-antiproteinase balance, nutritional status, and quality of life in stable chronic obstructive pulmonary disease due to tobacco and nontobacco etiology. Lung India. 2016 Nov-Dec;33(6):605-610. doi: 10.4103/0970-2113.192859. PMID 27890988